CLINICAL TRIAL: NCT01001143
Title: A Phase I Dose Escalation Study of Intravenous Decitabine in Combination With Oral Bexarotene in Patients With Acute Myeloid Leukemia (AML)
Brief Title: Intravenous (IV) Decitabine and Oral Bexarotene for Acute Myelogenous Leukemia (AML)
Acronym: AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-1661 / 201012801
Record Dates: First submitted 2009-10-19; First posted 2009-10-23 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Bexarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose Level 1 (Experimental): Decitabine 20 mg/m2 IV days 3-7 of cycle 1 and days 1-5 of subsequent cycles. Each cycle is 28 days.
  Bexarotene 100 mg/m2 PO daily for each 28 day cycle.
  Interventions: Drug: Decitabine; Drug: Bexarotene
- Dose Level 2 (Experimental): Decitabine 20 mg/m2 IV days 3-7 of cycle 1 and days 1-5 of subsequent cycles. Each cycle is 28 days.
  Bexarotene 200 mg/m2 PO daily for each 28 day cycle.
  Interventions: Drug: Decitabine; Drug: Bexarotene
- Dose Level 3 (Experimental): Decitabine 20 mg/m2 IV days 3-7 of cycle 1 and days 1-5 of subsequent cycles. Each cycle is 28 days.
  Bexarotene 300 mg/m2 PO daily for each 28 day cycle.
  Interventions: Drug: Decitabine; Drug: Bexarotene

INTERVENTIONS:
Drug: Decitabine
  Other Names: Dacogen®
Drug: Bexarotene
  Other Names: Targretin®

SUMMARY:
The main objective is to determine the safety and tolerability of combination decitabine and bexarotene during four cycles of therapy.

DETAILED DESCRIPTION:
The investigators are seeking to study the combination of decitabine and bexarotene. These two agents have each shown efficacy in decreasing leukemic blast counts and restoring normal hematopoiesis via different mechanisms of action and with non-overlapping side-effect profiles. By combining these agents, the investigators hope to improve overall response rates. The investigators further hope to improve platelet and neutrophil counts in an even greater number of patients, thus treating two of the most important sources of morbidity and mortality in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* AML with bone marrow blasts ≥ 20%.
* Relapsed disease after 1 or more lines of prior salvage chemotherapy and any FAB-AML, or
* Diagnosis of AML and age ≥ 60 and not a candidate for cytotoxic chemotherapy and any FAB-AML except FAB-M3.
* Performance status ≤ 2.
* Age ≥ 18 years.

Exclusion Criteria:

* Peripheral white blood cell count (WBC) > 10,000/microliter.
* Total bilirubin > 1.5 x normal.
* AST/ALT > 2.5 x normal.
* Serum creatinine > 2 x normal.
* Fasting serum triglyceride > 1,000 mg/dL.
* Active or poorly controlled graft vs host disease (GVHD).
* Pregnant or nursing.
* Known CNS leukemia.
* History of positive HIV serology.
* History of positive Hepatitis C serology.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, congestive heart failure of NYHA class 3 or 4, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.
* Chemotherapy within 21 days of enrollment.
* Radiation therapy within 14 days of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Toxicity of combination decitabine and bexarotene during four cycles of therapy | After 4 cycles of therapy

SECONDARY OUTCOMES:
To determine the complete remission (CR) and partial remission (PR) rate after four cycles of therapy. | After 4 cycles of therapy
To determine the rates of hematological improvement, transfusion independence, time to progression, cytogenetic response, and survival. | Every 2 months for 2 years after first dose of study drug
To perform correlative studies defining transcriptional response to bexarotene in primary AML bone marrow cells. | Baseline, C1D3, Day 25 of even cycles, and End of Study treatment
To perform correlative studies examining the clonality of morphologically differentiated neutrophils by fluorescence in situ hybridization (FISH) in patients with improved neutrophil counts. | Baseline, C1D3, Day 25 of even cycles, and End of Study treatment
To perform correlative studies comparing the self-renewal of morphologically differentiated neutrophils and leukemic blasts by colony forming assays in patients with improved neutrophil counts. | Baseline, C1D3, Day 25 of even cycles, and End of Study treatment
To perform correlative studies of platelet function by PFA100 in patients with platelet counts improved to >100,000/microliter | Baseline, C1D3, Day 25 of even cycles, and End of Study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Cashen, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu